CLINICAL TRIAL: NCT07020611
Title: Aneurysm SaC ManagemENt Device for Abdominal Aortic Aneurysms First-in-Human (ASCEND) Study
Brief Title: First-In-Human Study Evaluating Aneurysm Sac Lining in AAA Patients
Acronym: ASCEND
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Life Seal Vascular Inc. (Industry)
Collaborators: Auckland City Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP-0001
Record Dates: First submitted 2025-05-27; First posted 2025-06-13 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Abdominal Aortic Aneurysm
MeSH Terms: conditions — Aortic Aneurysm, Abdominal

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Cygnum ASMD Arm (Experimental)
  Interventions: Device: Cygnum Aneurysm Sac Management Device (ASMD)

INTERVENTIONS:
Device: Cygnum Aneurysm Sac Management Device (ASMD) — Cygnum ASMD, adjunctive to EVAR, lines the aneurysmal wall to prevent type II endoleaks

SUMMARY:
The goal of this clinical trial is to evaluate the safety and feasibility of the Cygnum Aneurysm Sac Management Device in patients with abdominal aortic aneurysms treated with endovascular aneurysm repair (EVAR). The main questions it aims to answer are:

1. Is the Cygnum device safe when used adjunctively with standard EVAR endografts?
2. Does it effectively reduce or prevent type II endoleaks by managing the aneurysm sac?

Participants will:

1. Undergo EVAR with adjunctive implantation of the Cygnum device
2. Have follow-up imaging (e.g., CT scans) and clinical assessments to evaluate device position and sac behavior over time

ELIGIBILITY:
Inclusion Criteria:

* Patient can understand the purpose of the trial, voluntarily participate in the trial and sign the informed consent
* Patient is willing to complete the follow-up according to the requirements of the protocol.
* Patient AAA anatomy complies with "instructions for use" for commercial EVAR devices used
* ≥18 years old
* Abdominal aortic aneurysm with sac diameter ≥ 5.5cm in males and ≥ 5.0cm in females
* Maximum blood flow luminal diameter ≤ 50mm
* Eligible for endovascular aneurysm repair based on anatomical considerations, such as adequate iliac/femoral access
* Patient is American Society of Anesthesiology (ASA) grade 1 through 3, inclusive.

Exclusion Criteria:

* Concomitant Common Iliac Artery aneurysms ≥ 25mm
* Life expectancy <2 years
* Already participating in an investigational drug or device study
* Known allergy or contraindication to any study device material
* Coagulopathy or uncontrolled bleeding disorder
* Ruptured, leaking, inflammatory or mycotic aneurysm
* Connective tissue diseases (e.g., Marfan Syndrome)
* Unsuitable vascular anatomy that may interfere with device introduction or deployment, in the opinion of the investigator
* Aneurysmal or dissected disease of the descending thoracic aorta
* Previous surgical or EVAR repair for AAA
* Myocardial infarction and/or major heart surgery ≤ 90 days prior to the procedure
* Transient Ischemic Attack or stroke ≤ 90 days prior to the procedure
* Unstable angina or other active cardiac condition such as congestive heart failure, untreated or worsening atrial arrhythmia, ventricular arrhythmia or valvular disease ≤ 30 days prior to the procedure
* Unable or unwilling to comply with study follow-up requirements
* Serum creatinine level ≥ 180 µmol/L
* Patients of childbearing potential who are pregnant or planning to become pregnant during the course of the study
* Patient has other medical, social or psychological problems that, in the opinion of the investigator, study involvement would not be in their best interest.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-11-26 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Incidence of major adverse events (MAEs) | 30 days post-procedure
  Rate of related major adverse events (MAEs)
Procedural Technical Success | Immediately after the intervention
  Technical success, defined as lining the AAA sac wall with the investigational devices

SECONDARY OUTCOMES:
Incidence of related major adverse events (MAEs) | 12 months post procedure
  Incidence rate of related major adverse events (MAEs)
Incidence of related serious adverse events (SAEs) | 12 months post procedure
  Incidence rate of related serious adverse events (SAEs)
Efficacy - Type II endoleaks | 12 months post procedure
  Incidence of type II endoleaks
Efficacy - AAA sac diameter | 12 months post procedure
  Change in AAA sac diameter

CONTACTS AND LOCATIONS:
Overall Officials: Raja Ghanem, Study Director — Life Seal Vascular Inc.
Locations (1):
- Auckland City Hospital, Auckland, New Zealand

IPD SHARING:
Plan to Share IPD: No